CLINICAL TRIAL: NCT06797388
Title: The Effect of Thyroid Lobe Volume on the Common Carotid Artery Blood Flow in Thyroidectomy Position
Brief Title: The Effect of Thyroid Lobe Volume on the Common Carotid Artery Blood Flow
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Başar Erdivanlı, Assoc. Prof., Recep Tayyip Erdogan University
Other Study IDs: 2016/21
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Surgery; Head Extension on the Anatomic Axes of the Superior Airway
Keywords: common carotid artery; common carotid artery blood flow; Doppler ultrasonography; thyroid volume; cerebral oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Normal size: Right or left side of any patient with a normal thyroid lobe size according to gender-specific limits of normal thyroid volume (15 ml for adult females, 18 ml for adult males)
- Large size: Right or left side of any patient with a large thyroid lobe size according to gender-specific limits of normal thyroid volume (15 ml for adult females, 18 ml for adult males)

SUMMARY:
The goal of this observational study is to evaluate how thyroid lobe volume affects carotid artery blood flow dynamics in adult patients undergoing elective thyroidectomy. The study includes male and female participants aged 18 years and older who have euthyroid function and are scheduled for elective thyroidectomy.

The main questions it aims to answer are:

* Does thyroid lobe volume influence carotid artery blood flow characteristics, particularly systolic/diastolic flow time ratios, during thyroidectomy?
* What is the optimal thyroid lobe volume cutoff for predicting altered systolic/diastolic flow time ratios (<0.3)?

Participants will:

* Undergo Doppler ultrasound measurements at three time points: before anesthesia induction, after anesthesia induction, and after surgical positioning.
* Have their carotid artery blood flow and regional cerebral oxygenation values assessed.

No comparison groups are involved, as all participants will be observed under the same conditions.

DETAILED DESCRIPTION:
This observational study investigates how the size of the thyroid gland affects blood flow in the common carotid artery during thyroidectomy, a surgical procedure to remove part or all of the thyroid gland. The thyroid gland is anatomically close to the carotid artery, a major blood vessel supplying blood to the brain. Enlarged thyroid lobes may compress the artery, potentially altering blood flow dynamics, particularly during the semi-Fowler's position required for the surgery. By examining these effects, this study aims to provide insights into the interplay between thyroid anatomy and carotid blood flow, which could have implications for surgical and anesthetic management.

Study Objectives

The primary objective is to determine the relationship between thyroid lobe volume and carotid artery blood flow during thyroidectomy. Specifically, the study seeks to:

1. Evaluate how thyroid lobe volume influences systolic and diastolic blood flow in the carotid artery.
2. Identify a thyroid lobe volume cutoff associated with significant alterations in systolic/diastolic flow time ratios (<0.3).

Study Population

The study includes adult patients aged 18 years and older scheduled for elective thyroidectomy. Participants must be in a euthyroid state, as thyroid hormone abnormalities may influence recovery and perioperative outcomes. Patients with conditions such as anemia, labile hypertension, or prior thyroid surgeries, as well as pregnant or emergency cases, are excluded.

Study Design

This is a prospective observational study conducted at a tertiary academic hospital. Measurements are obtained from each participant at three critical time points:

1. Baseline (T0): Before anesthesia induction.
2. After anesthesia induction (T1).
3. After surgical positioning (T2): In the semi-Fowler's position with head extension.

Doppler ultrasound is used to assess carotid artery diameters and flow velocities. Regional cerebral oxygenation is also measured using a cerebral oximeter to evaluate the impact of altered blood flow on brain perfusion.

Study Methods

Participants undergo the following procedures during the study:

* Ultrasound Measurements: The diameters of the common carotid artery at systole and diastole are measured, and Doppler flow velocities (peak systolic velocity, end-diastolic velocity) are recorded. These values are used to calculate mean velocity, Gosling pulsatility index, and Pourcelot resistance index.
* Manual Tracing of VTI: In cases with altered systolic/diastolic flow ratios, manual tracing is used to ensure accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) scheduled for elective thyroidectomy.
* Patients in a euthyroid state as confirmed by recent laboratory tests.
* Ability to provide written informed consent.

Exclusion Criteria:

* Pregnant patients.
* Emergency thyroidectomy cases.
* History of subtotal thyroidectomy.
* History of allergic reaction to anesthetic agents.
* Presence of anemia (hemoglobin levels below local institutional thresholds).
* Presence of labile hypertension (documented by repeated measurements on the surgical ward)
* Presence of abnormal thyroid hormone levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients scheduled for elective thyroidectomy at a tertiary academic hospital. Participants are drawn from the hospital's general surgery clinic, which serves a diverse population from both urban and surrounding rural areas. Patients undergoing surgery for various thyroid pathologies, including benign nodules and malign pathologies, are included. All participants are assessed preoperatively to ensure they meet the study's inclusion criteria, including euthyroid status, and are representative of individuals typically undergoing elective thyroid surgery in this clinical setting.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Change in Systolic/Diastolic Flow Time Ratio of the Common Carotid Artery | Measured at baseline (T0), post-anesthesia induction (T1), and post-surgical positioning (T2).
  Assess the relationship between thyroid lobe volume and alterations in the systolic/diastolic flow time ratio during thyroidectomy.
Thyroid Lobe Volume Cutoff for Altered Flow Dynamics | Post-hoc analysis using data from baseline (T0).
  Determine the thyroid lobe volume cutoff associated with a systolic/diastolic flow time ratio <0.3.

SECONDARY OUTCOMES:
Change in Carotid Artery Blood Flow | Measured at baseline (T0), post-anesthesia induction (T1), and post-surgical positioning (T2).
  Evaluate how thyroid lobe volume affects carotid artery blood flow during different surgical time points.
Regional Cerebral Oxygenation Changes | Measured at baseline (T0), post-anesthesia induction (T1), and post-surgical positioning (T2).
  Measure the impact of altered carotid artery blood flow on regional cerebral oxygenation during thyroidectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Başar Erdivanlı, Assoc. Prof., Study Director — Recep Tayyip Erdogan University Medical Faculty
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The raw data supporting the reported results and the R source files used during the analysis will be made available by the authors on reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The individual participant data (IPD) and supporting information, including the study protocol, statistical analysis plan, and analytic code, will be available starting 6 months after publication of the study results. Data will remain available indefinitely for academic purposes.
Access Criteria: Access to the IPD and supporting information will be provided upon reasonable request to researchers affiliated with academic institutions. Requestors must provide proof of academic affiliation and a clear statement of their intended use of the data. Requests will be reviewed by the corresponding author to ensure alignment with the study's objectives and ethical considerations. Data will be shared through secure data transfer mechanisms.

REFERENCES:
- [Background] Braakman HM, Knippenberg SA, de Bondt BJ, Lodder J. An unusual cause of transient neurologic deficits: compression of the carotid artery by a thyroid cystic nodule. J Stroke Cerebrovasc Dis. 2010 Jan;19(1):73-4. doi: 10.1016/j.jstrokecerebrovasdis.2009.02.007. PMID 20123230
- [Background] Saracoglu A, Altun D, Yavru A, Aksakal N, Sormaz IC, Camci E. Effects of Head Position on Cerebral Oxygenation and Blood Flow Velocity During Thyroidectomy. Turk J Anaesthesiol Reanim. 2016 Oct;44(5):241-246. doi: 10.5152/TJAR.2016.77598. Epub 2016 Oct 1. PMID 27909604